CLINICAL TRIAL: NCT05888974
Title: Diagnostic Performance of the Mitral Annulus Velocity Variation Measured by Tissue Doppler to Evaluate the Fluid Responsiveness During the Initial Management of Shock in Patients Admitted to the Emergency Department
Acronym: EVO-E'
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-A00022-43
Record Dates: First submitted 2023-05-25; First posted 2023-06-05 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Shock
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with shock (MAP < 65 mmHg) requiring vascular filling: The study population consisted of patients with shock (MAP < 65 mmHg) requiring vascular filling indicated by the referring physician physician, recruited consecutively in the emergency department of the CHU of Nîmes and Montpellier.
  Interventions: Diagnostic Test: Cardiac ultrasonography

INTERVENTIONS:
Diagnostic Test: Cardiac ultrasonography — During the inclusion visit, the patient will receive 3 cardiac ultrasonography. The first one will be performed at the time of the initiation of the 500mL vascular filling (T0), without delaying and the second one after the end of the filling (Tfin). These first two ultrasound are part of standard practice. A third will be performed 20 minutes after the end of the vascular filling (Tfin+20).

SUMMARY:
Assessing the response to vascular filling in shock is a challenge in emergency medicine.

The mitral annulus velocity measured by tissue Doppler (E') has recently been characterized as sensitive to the preload conditions of a patient.

The investigators hypothesize that the E' variation (∆E') before and after fluid filling allows us to assess the response to vascular filling. The investigators hypothesize that the ∆E' has a good diagnostic performance to establish whether a patient is responsive to fluid filling, defined by an area under the ROC curve greater than 0.75.

DETAILED DESCRIPTION:
Assessing the response to vascular filling in shock is a challenge in emergency medicine.

Trans thoracic ultrasound (TTS) is recommended for the diagnosis and management of this type of patient. TTS allows real-time monitoring of the effectiveness of a therapeutic . In case of circulatory failure without cardiac failure, it is recommended to perform fluid filling tests based on an increase in of indicators to assess preload dependence. The change in subaortic VTI, which has become the gold standard in clinical practice for diagnosing fluid filling response, suffers from a lack of technical feasibility. The mitral annulus velocity measured by tissue Doppler (E') has recently been characterized as sensitive to the preload conditions of a patient. The high feasibility of this technique makes its study interesting for the evaluation of the preload (and its variation after variation after vascular filling) of the patient in shock in the emergency department. To our knowledge, there are no clinical studies exploring the relevance of this technique to evaluate fluid filling response in patient admitted with shock in the emergency department.

The investigators hypothesize that the E' variation (∆E') before and after fluid filling allows us to assess the response to vascular filling. The investigators hypothesize that the ∆E' has a good diagnostic performance to establish whether a patient is responsive to fluid filling, defined by an area under the ROC curve greater than 0.75.

The main objective of this study is to investigate the diagnostic performance of ∆E' in establishing response to fluid filling in a prospective cohort of patients admitted to the emergency department with shock requiring vascular filling.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been informed of the study and does not refuse to participate.
* Patient is at least ≥ 18 years of age.
* The patient must be beneficiary of a health insurance plan.
* Patient has shock with a mean blood pressure less than 65 mmHg (<)
* The patient does not have acute intracranial pathology
* The referring physician has decided on a vascular filling with 500mL of crystalloids (NaCl 0.9% or Ringer lactate)

Exclusion Criteria:

* The patient has already received 2 vascular fillings since the beginning of his management
* The patient is in shock and has a contraindication to vascular filling : shock of a cardiogenic or obstructive nature
* The patient has an intracranial pathology requiring maintain a MAP ≥ 80 mmHg
* The patient is intubated or on Non-Invasive Ventilation before the vascular filling
* The patient is under court protection
* The patient is pregnant, parturient or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consisted of patients with shock (MAP < 65 mmHg) requiring vascular filling indicated by the referring physician physician, recruited consecutively in the emergency department of the CHU of Nîmes and Montpellier.
Sampling Method: Non-Probability Sample
Enrollment: 187 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-08-08 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
E' variation (∆E') | Inclusion time
  The E' wave will be measured by tissue Doppler at the initiation (T0) of the filling and after the end of the vascular (Tfin) to determine its variation (%) between these two times of measurement.
Fluid filling responsiveness | Inclusion time
  Vascular filling is defined by the intravenous administration of 500 mL of crystalloid for 20 to 30 minutes, decided by the physician in charge. The response to filling will be evaluated by the variation of the time velocity index between T0 and Tfin (∆ITV) measured with pulsed Doppler.
  Patients will be considered :
  * Responder (R) group if ∆ITV ≥ 15%
  * Nonresponder group (NR) if ∆ITV < 15%.

SECONDARY OUTCOMES:
∆E'late | Inclusion time
  ∆E'late: the E' wave will be measured by trans thoracic ultrasound before vascular filling (T0) and 20 minutes after the end of vascular filling (Tfin+20) to determine its variation (%) between these two times of measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nîmes, Nîmes, France

IPD SHARING:
Plan to Share IPD: Undecided